CLINICAL TRIAL: NCT05488288
Title: Bariatric Surgery With Mesh Repair of Ventral Hernia: a Randomized Controlled Trial
Acronym: BeSURE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP211049; 2023-A00658-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-07-28; First posted 2022-08-04 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Ventral Hernia
Keywords: Ventral Hernia; Bariatric surgery; Obesity; Mesh repair; Suture
MeSH Terms: conditions — Hernia, Ventral; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh group (Experimental): ventral hernia repair with non absorbable mesh placement concomitant to bariatric procedure (sleeve gastrectomy or by-pass).
  In this group, the repair technique and the type of mesh are left to the choice of the center, as there are no strong data to demonstrate which technique is the best for VH repair in this population.
  Interventions: Procedure: Mesh repair
- Suture group (Active Comparator): suture repair of ventral hernia concomitant to bariatric procedure (sleeve gastrectomy or by-pass).
  In this group, the hernia sack is resected through an open approach, and the fascial defect is systematically closed with a slowly absorbable monofilament suture.
  Interventions: Procedure: Suture repair

INTERVENTIONS:
Procedure: Mesh repair — Abdominal ventral hernia (VH) repair with mesh during bariatric surgery. the repair technique and the type of mesh are left to the choice of the center, as there are no strong data to demonstrate which technique is the best for VH repair in this population.
  Arms: Mesh group
Procedure: Suture repair — The hernia sack is resected through an open approach, and the fascial defect is systematically closed with a slowly absorbable monofilament suture.
  Arms: Suture group

SUMMARY:
The primary objective of the study is to demonstrate that hernia recurrence (VH) repair with non absorbable mesh concomitant to Bariatric Surgery (BS) decreases the risk of VH, with or without surgical repair, during the first two years after BS when compared to VH suture repair without mesh.

As secondary objectives, the study aims to assess the impact of concomitant VH repair with non absorbable mesh versus suture repair in morbidly obese BS candidates on the following measures: - hernia recurrence at 1 year after randomization; - reoperation for hernia recurrence at 2 years after randomization; - strangulated hernia, surgical infection and mesh bulging at one year after randomization; - postoperative morbidity and mortality at 90 days after randomization; - benefit-risk ratio; - chronic pain at three months, six months, one year and two years after randomization; - quality of life during the two years after randomization; - incremental cost utility ratio; - short- and mid-term weight loss. To study if the efficacy of mesh versus suture VH repair differs according to the type and size of VH and to the surgical technique.

DETAILED DESCRIPTION:
This is a prospective, multicentric, superiority, comparative randomized (1:1) single-blinded clinical trial with blinded assessment of the primary endpoint.

Hypothesis for the study: abdominal ventral hernia (VH) repair with mesh during bariatric surgery (BS) is more effective than suture repair in preventing VH recurrence. Secondarily, we expect that mesh repair would not increase the risk of surgical site infection.

Population of study participants:

Patients between 18 and 60 years, presenting with VH and scheduled for BS, excluding pregnant women and protected adults.

All consecutive eligible patients will be invited to participate by visceral surgeons during preoperative consultations for BS. Included patients will be randomly assigned (1/1 ratio) to either mesh VH repair (intervention group) or suture VH repair (control group) by visceral surgeons at hospital admission (hospitalization or outpatient surgery) for BS and VH repair.

Patients will be followed according to clinical guidelines for BS follow-up at M1, M3, M6, M9, M12, M18 and M24 after BS.

There will be 29 surgical centers in France (digestive surgeons), targetting 354 eligible patients.

Statistical analysis:

An intention-to-treat statistical analysis will be performed at the end of the follow-up, when primary endpoint of all randomized patients will be documented.

The analysis for the primary endpoint will consist in comparing proportions of hernia recurrence during the two years after surgery between the two arms, using a Chi2 test.

An interim analysis is planned after half of the subjects finished their follow-up, in order to confirm the efficacy of the intervention arm, or alternatively its lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years.
* Body Mass Index (BMI) ≥ 40 kg/m² or ≥ 35 kg/m² associated with at least one comorbidity that can improve after BS.
* Body Mass Index (BMI) < 50 kg/m².
* Primary or first recurrent incisional midline VH, umbilical or epigastric, width between 1 cm and 4 cm, on abdominopelvic CT-scan without contrast injection.
* Decision for primary sleeve gastrectomy or by-pass after multidisciplinary discussion.
* Request for BS approved by health insurance authorities.
* Written informed consent from patient.

Exclusion Criteria:

* Previous VH repair with mesh.
* Other types of abdominal hernia (lateral, subxiphoidal, infraumbilical, suprapubic, parastomal, non-midline port-site, and groin hernia).
* Decision of performing BS by laparotomy.
* Reoperation for BS (excepted previous adjustable gastric banding).
* Ongoing abdominal skin infection.
* Emergency surgery.
* ASA (American Society of Anesthesiologists) score>3.
* Ongoing pregnancy or breast-feeding.
* Patient not covered by social insurance.
* Patient under legal guardianship.
* Patient already included in a clinical trial on hernia recurrence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence rate, with or without surgical repair | at 2 years
  Final diagnosis of hernia recurrence will be made by an endpoint committee of radiologists, blinded to the randomization arm (it is not possible to distinguish mesh from suture repair on CT-scans) on abdomino-pelvic CT-scan without contrast injection.
  Radiological hernia is defined as any protrusion of abdominal contents, including the anterior parietal peritoneum, visible as discontinuity of the fascial layers.
  In case of hernia recurrence requiring new VH repair during the study period (before the two years CT-scan evaluation), this will be considered as an event in intention-to-treat analysis.

SECONDARY OUTCOMES:
Hernia recurrence rate at 1 year | at 1 year
  Hernia recurrence rate clinically
Reoperation rate for recurrence at 2 years | at 2 years
  Reoperation rate for recurrence, at 2 years after randomization with medical files.
Strangulated hernia rate at 1 year | at 1 year
  Strangulated hernia rate (requiring emergent surgery), at 1 year after randomization (medical files)
Surgical site infection rate at 1 year | at 1 year
  Surgical site infection rate (superficial or deep), at 1 year after randomization (medical files)
Mesh bulging rate at 2 years | at 2 years
  Mesh bulging rate, defined by a protrusion of the mesh through a fascial defect without hernia recurrence at CT-scan evaluation, at 2 years after randomization.
Postoperative morbidity rate | daily up to 90 days
  Postoperative morbidity rate (any complication in the 90 days after randomization).
Postoperative mortality rate | daily up to 90 days
  Postoperative mortality rate (any complication in the 90 days after randomization).
Benefit-risk ratio | at the end of the study
  Benefit-risk ratio (DOOR-RADAR score established by the scientific committee prior to the start of the study).
Self-reported chronic pain | at 3 months, 6 months, 1 year and 2 years
  Self-reported chronic pain, using the Visual Analogue Scale, at 3 months, 6 months, 1 year and 2 years after randomization
Score of quality of life | at 3 months, 6 months, 1 year and 2 years
  Using the EQ-5D-5L self-questionnaire EuroQol-5Dimensions-5Levels self-questionnaire (EQ-5D-5L value : -0.530 to 1.0 ; 1.0 indicates the best quality of life)
Pain evaluation | at 3 months, 6 months, 1 year and 2 years
  Using Visual Analogue Scale Visual Analogue Scale (0 to100; 0 represents 'no pain at all' whereas 100 represents 'the worst pain ever possible')
Incremental cost utility ratio | at 2 years
  Cost will be calculated.
Weight loss | at 3 months, 6 months, 1 year and 2 years
  Short-term weight loss (percentage of excess weight loss at 3 and 6 months after the procedure); mid-term weight loss (percentage of excess weight loss at 1 and 2 years after the procedure).
Hernia recurrence rate at 2 years | at 2 years
  Hernia recurrence rate at 2 years after randomization, by type (primary or incisional) and size of VH and by surgical technique (sublay/retromuscular or intraperitoneal or preperitoneal/underlay).

CONTACTS AND LOCATIONS:
Overall Officials: David MOSZKOWICZ, MD, PhD, Principal Investigator — Department of visceral and digestive surgery, Louis-Mourier hospital, APHP
Locations (1):
- Department of visceral and digestive surgery, Louis Mourier hospital, APHP, Colombes, France